CLINICAL TRIAL: NCT02693496
Title: Mobile Lung Nodule Observatory for Worldwide, Evidenced - Based Research
Brief Title: Mobile Lung Nodule Observatory for Worldwide, Evidenced-based Research
Acronym: mLOWER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Alliance Against Lung Cancer (Other)
Responsible Party: Principal Investigator, Bai Chunxue, Professor, Chinese Alliance Against Lung Cancer
Other Study IDs: CAALC-002-mLOWER
Record Dates: First submitted 2015-10-27; First posted 2016-02-26 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Solitary Pulmonary Nodule
Keywords: ResearchKit; CT screening; Early Diagnosis; Lung Cancer
MeSH Terms: conditions — Solitary Pulmonary Nodule; Disease; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Installation or registration of smartphone application — Completed the installation and registration of mobile terminal software online

SUMMARY:
Patients with lung nodules may develop a variety of potentially severe symptoms. These symptoms may impact a patient's quality of life and lead to difficult treatment. Through this research program, the investigators want to understand the pathogenesis of the changes of these symptoms.

DETAILED DESCRIPTION:
Lung nodules can manifest as single or multiple independent lung consolidation shadow in form of quasi-circular. These lung nodules are surrounded by normal lung tissues, and will not cause pulmonary atelectasis. In some early standards, all the quasi-circular shadows within 6cm found in lung are categorized as lung nodules. However, according to current standards, the lesion within 3cm can be identified as lung nodules. With widespread use of lung cancer CT screening, lung nodules were identified more and more frequently.

What is the optimal way to manage this CT finding? Should we adopt surgical removal or just observation? An optimal solution is to determine a clearly defined standard of care that is easy to learn. We propose a method called "three plus two". The 'Three' is a three-step testing method, and the 'Two' means two alternative solutions. Three-step testing method includes collecting medical history, non-invasive examination, and invasive examination. The two alternative solutions are surgical removal and follow-up observation. We have independently developed an application based on a smartphone platform. This platform will provide a novel evidence-based research method for observing the dynamic evolution of the lung nodules in patients. There have been no prior studies about managing this CT scan finding, either in China or internationally.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90
* There is a chest lesion less than 3cm width (examined by Thin-Section CT)
* The patient or his family member owns a smartphone
* Signed informed consent
* Completed the installation and registration of mobile terminal software online
* Willing to complete a 10-year period of follow-up

Exclusion Criteria:

* Not equipped with a smartphone
* Cannot complete the installation or registration of smartphone application software online
* Received prior chemotherapy medications for lung cancer or received lung surgical removal treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 10,000 patients will participate in this research program, in 100 different medical institutions.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-10; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic accuracy among different type of lung nodules. | 10 years
  Utilizing the professional statistical software (SPSS 15.0), through T-test, Mann-Whitney U test, and analyzing the receiver operating characteristic (ROC) curve, to compare the diagnostic accuracy among different type of lung nodules. A p<0.05 cutoff will be the standard used to determine statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, M.D, Ph.D, Study Chair — Chinese Alliance Against Lung Cancer
Locations (34):
- China (34):
  - Beijing Union Hospital, Beijing
  - General Hospital of PLA, Beijing
  - Hebei Pronvince Cangzhou City People's Hospital, Cangzhou
  - Xiaya Hospital Central South Unversity, Changsha
  - Anhui Province Chaoyang Hospital, Chaoyang
  - West China Hospital Sichuan University, Chengdu
  - No.1 Hospital Chongqing Medical University, Chongqing
  - Western East Hospital No. 3 PLA Medical University, Chongqing
  - No. 2 Hospital Dalian Medical University, Dalian
  - Guizhou Province People's Hospital, Guizhou
  - International Hospital Zhejiang University, Hangzhou
  - No. 1 Hospital Zhejiang University Medical College, Hangzhou
  - Yunnan Province Cancer Hospital, Kunming
  - Shandong Province Liaocheng City People's Hospital, Liaocheng
  - No. 2 Hospital Fujian Medical University, Quanzhou
  - Kecheng District Hospital, Quzhou
  - Shanghai Zhongshan Hospital, Shanghai
  - Minhang District Hospital Fudan University, Shanghai
  - Putuo District Central Hospital Shanghai Chinese Medical University, Shanghai
  - Ruici Clinic, Shanghai
  - No. 2 Hospital Tianjin Chinese Medical University, Tianjin
  - Weifang City No.2 People's Hospital, Weifang
  - Wudang Hospital Guiyang Medical College, Wudang
  - Wuhu City No. 2 Hopsital, Wuhu
  - No. 5 Wuxi People's Hospital, Wuxi
  - Xining Hospital No.4 PLA University, Xi'an
  - Xiamen City No.3 People's Hospital, Xiamen
  - Yantai City Taishan Hopsital, Yantai
  - Henan Province People's Hospital, Zhengzhou
  - No. 1 Hospital Zhengzhou University, Zhengzhou
  - Shandong Pronvince Zibo City Official Hospital, Zibo
  - Shandong Province Linzi District Hospital, Zibo
  - Sichuan Province Zigong City No. 1 Hospital, Zigong
  - Guizhou Province Zunyi Medical College Hospital, Zunyi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang DW, Zhang Y, Hong QY, Hu J, Li C, Pan BS, Wang Q, Ding FH, Ou JX, Liu FL, Zhang D, Zhou JB, Song YL, Bai CX. Role of a serum-based biomarker panel in the early diagnosis of lung cancer for a cohort of high-risk patients. Cancer. 2015 Sep 1;121 Suppl 17:3113-21. doi: 10.1002/cncr.29551. PMID 26331818
- [Background] Gould MK, Donington J, Lynch WR, Mazzone PJ, Midthun DE, Naidich DP, Wiener RS. Evaluation of individuals with pulmonary nodules: when is it lung cancer? Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e93S-e120S. doi: 10.1378/chest.12-2351. PMID 23649456